CLINICAL TRIAL: NCT04006665
Title: Role of Lung Ultrasonography in Diagnosing Atelectasis in Robotic Pelvic Surgeries
Acronym: Lung US
Status: Completed | Type: Observational
Sponsor: Rajiv Gandhi Cancer Institute & Research Center, India (Other)
Responsible Party: Principal Investigator, Dr Anita Kulkarni, Principal Investigator, Rajiv Gandhi Cancer Institute & Research Center, India
Other Study IDs: RGCIRC Lung US
Record Dates: First submitted 2019-05-02; First posted 2019-07-05 (Actual); Last update posted 2023-04-21 (Actual); Status verified 2023-04

CONDITIONS: Atelectasis
Keywords: Lung Ultrasonography; Step Trendelenburg position
MeSH Terms: conditions — Pulmonary Atelectasis

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Lung Ultrasonography prior to docking Robotic arms: Base line Lung ultrasonography will be performed in three basal zones for Right and Left lung -Post intubation and prior to docking robotic arms .
  Interventions: Diagnostic Test: Lung Ultrasonography (Baseline)
- Lung Ultrasonography after removal of robotic arms: Lung Ultrasonography will be performed to assess degree of atelectasis after removal of robotic arms and before extubation in three basal zones for Right and Left lung .
  Interventions: Diagnostic Test: Lung Ultrasonography ( At the end of surgery)

INTERVENTIONS:
Diagnostic Test: Lung Ultrasonography (Baseline) — Lung Ultrasonography will be performed prior to docking Robotic arms in basal three lung zones on both sides.
  Groups: Lung Ultrasonography prior to docking Robotic arms
Diagnostic Test: Lung Ultrasonography ( At the end of surgery) — Lung Ultrasonography will be performed after removal of Robotic arms and before extubation in basal three lung zones on both sides to assess degree of atelectasis.
  Groups: Lung Ultrasonography after removal of robotic arms

SUMMARY:
General anaesthesia results in developement of atelectasis in dependent areas of the lungs exposing patients to an increased risk of hypoxaemia.During pelvic robotic surgeries pneumoperitoneum and steep trendelenburg position further increases atelectasis. Lung Ultrasound imaging is a promising , noninvasive , non-radiant, portable tool to study intraoperative lung atelectasis.

DETAILED DESCRIPTION:
Methodology -In the Operation Room 5 lead Electrocardiogram (ECG) , Pulse Oximetry (SPO2 ) , Noninvasive blood pressure (NIBP), End tidal carbon di Oxide (ETCO2 )and core temperature will be monitored , intravenous assess will be established with large bore cannula ,under Local anesthesia Radial artery cannulation will be performed , standard general anesthesia with oral cuffed Endotracheal tube and Intermittent Positive Pressure Ventilation (IPPV ) will be provided to all patients.Anaesthesia will be induced with Fentanyl 1-2 mcg/kg-1 , Morphine 0.5mg/kg-1 ,Propofol sleeping dose , Atracurium 0.5mg/kg-1,and maintained with Air/O2 Sevoflurane , Propofol infusion @100- 150 mcg/kg-1 to maintain Bispectral Index (BIS) between 40 -60 and atracurium infusion to maintain Train -of - Four (TOF Ratio) < 0.5 Baseline Lung Ultrasound Imaging will be performed to record 4 point Lung aeration score ( 0= Normal lung /No aeration loss , 1= mild aeration loss, 2=moderate aeration loss ,3=severe aeration loss ) at T1 - 5 minutes after induction of anaesthesia and before docking robotic instruments in 6 basal zones in both lungs ( 3 zones in each lung ) and labelled as Zone I (Right anterior basal ) Zone II ( Right lateral basal) and Zone III (Right posterior basal) . Zone IV ( Left anterior basal) , Zone V (Left lateral basal ) , Zone VI ( Left Posterior basal ).T2 - Lung Ultrasound Imaging will be performed to record aeration score after removal of robotic arms at the end of robotic surgery and before extubation in 6 basal zones in both lungs.Ti Arterial blood gas 5 minutes after induction of anesthesia and before docking robotic instruments.Tii -Arterial blood gas 5 minutes after the end of robotic surgery and de docking robotic instruments.All patients will receive Positive End Expiratory Pressure (PEEP) 5 cms of water (H2O) intraoperatively . Intraabdominal Pressure will be maintained at 15 cms H2O. Any decrease in Oxygen saturation < 96 % and intervention required will be noted. At the end of surgery , neuromuscular blockade will be reversed , trachea extubated and patient shifted to Postanaesthesia Care Unit.

ELIGIBILITY:
Inclusion Criteria:

* Patients undergoing Robotic Pelvic surgeries under general anaesthesia

Exclusion Criteria:

* Lung consolidation
* Lung fibrosis
* Cardiac failure
* Previous thoracic surgery
* BMI > 32

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients undergoing pelvic robotic surgery under general anaesthesia.
Sampling Method: Non-Probability Sample
Enrollment: 50 (Actual)
Dates: Start 2019-09-01 (Actual); Primary Completion 2020-02-19 (Actual); Study Completion 2020-02-28 (Actual)

PRIMARY OUTCOMES:
To assess the degree of lung atelectasis and aeration score. | T1 -Baseline postintubation and before docking robotic arms .T2 - At the end of Robotic surgery upto 6 hours and after removal of robotic arms before extubation.
  By performing Lung Ultrasonography in six basal zones ( 3 in each lung)

SECONDARY OUTCOMES:
To study the effect of intraoperative Atelectasis on arterial oxygen tension | T1 - Baseline postintubation and before docking robotic arms , T2 -upto 6 hours of robotic surgery and after removal of robotic arms ..
  Arterial Oxygen tension (PaO2) in mmHg
To study the effect of intraoperative atelectasis on Alveolar- arterial Oxygen Gradient | T1 - Baseline postintubation and before docking robotic arms , T2 -upto 6 hours of robotic surgery and removal of robotic arms before extubation.
  Alveolar - arterial Oxygen gradient will be obtained .
To study the effect of mode of ventilation on intraoperative atelectasis | T1 Baseline T2 Upto 6 hours of Robotic surgery
  Volume controlled ventilation and pressure controlled ventilation if peak airway pressure exceed 35

CONTACTS AND LOCATIONS:
Overall Officials: Anita Kulkarni, M.D., Principal Investigator — RajivGandhi Cancer Institute and Research centre , Delhi ,India
Locations (1):
- Rajiv Gandhi Cancer Institute and Research Centre, Delhi, India

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Acosta CM, Maidana GA, Jacovitti D, Belaunzaran A, Cereceda S, Rae E, Molina A, Gonorazky S, Bohm SH, Tusman G. Accuracy of transthoracic lung ultrasound for diagnosing anesthesia-induced atelectasis in children. Anesthesiology. 2014 Jun;120(6):1370-9. doi: 10.1097/ALN.0000000000000231. PMID 24662376